CLINICAL TRIAL: NCT01662674
Title: A Randomized, Open-label, Oral Single Dosing, Two-way Crossover Clinical Trial to Compare the Safety/Tolerability and Pharmacokinetics/Pharmacodynamics of the Combinations of Gemigliptin 50mg and Metformin HCl Extended Release 1000mg in Comparison to Each Component Administered in Healthy Male Volunteers
Brief Title: BE Study of the Combinations of Gemigliptin 50mg and Metformin HCl Extended Release 1000mg in Comparison to Each Component Administered Alone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LG-DMCL002
Record Dates: First submitted 2012-08-06; First posted 2012-08-10 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
MeSH Terms: interventions — LC15-0444

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- G+M (Experimental): Coadministration of gemigliptin 50mg and metformin HCl extended release 1000mg
  Interventions: Drug: gemigliptin and metformin HCl extended release
- C (Experimental): Combination of gemigliptin50mg/metformin HCl extended release 1000mg
  Interventions: Drug: gemigliptin/metformin HCl extended release

INTERVENTIONS:
Drug: gemigliptin and metformin HCl extended release — Coadministration of gemigliptin 50mg and metformin HCl extended release 1000mg, for 1 day
  Arms: G+M
Drug: gemigliptin/metformin HCl extended release — Administration of combination of gemigliptin 50mg/metformin HCl extended release 500mg, for 1day.
  Arms: C

SUMMARY:
This study is to evaluate the safety/tolerability and pharmacokinetics/pharmacodynamics of the combinations of gemigliptin 50mg and metformin HCl extended release 1000mg in comparison to each component administered in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 to 45, healthy male subjects(at screening)
* Body weight between 55kg - 90kg, BMI between 18.0 - 27.0
* FPG 70-125mg/dL glucose level(at screening)
* Subject who totally understand the progress of this clinical trials, make decision by his free will, and signed a consent form to follow the progress.

Exclusion Criteria:

* Subject who has past or present history of any diseases following below.(liver including hepatitis virus carrier, kidney, Neurology,immunology,pulmonary,endocrine,hematooncology,cardiology,mental disorder.)
* Subject who had GI tract disease or(ulcer, acute or chronic pancreatitis) surgery.(appendectomy, hernioplasty are not included)
* Subject who had drug hypersensitivity reaction.(Aspirin, antibiotics)
* Subject who already participated in other trials in 3months
* Subject who had whole blood donation in 2months, or component blood donation in 1months or transfusion in 1months currently.
* Smokers.(but, if the subject did'nt smoke in 3months, can participate the trial)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2012-10; Primary Completion 2012-11 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
AUClast | up to 48h post-dose
  To evaluate AUClast of gemigliptin and metformin
Cmax | up to 48h post-dose
  To evaluate Cmax of gemigliptin and metformin

SECONDARY OUTCOMES:
AUEC | up to 48h post-dose
  This parameter is been used to measure pharmarcodynamic characters of gemigliptin and metformin, the supression rate of DPP4 activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Park SI, Lee H, Oh J, Lim KS, Jang IJ, Kim JA, Jung JH, Yu KS. A fixed-dose combination tablet of gemigliptin and metformin sustained release has comparable pharmacodynamic, pharmacokinetic, and tolerability profiles to separate tablets in healthy subjects. Drug Des Devel Ther. 2015 Feb 4;9:729-36. doi: 10.2147/DDDT.S75980. eCollection 2015. PMID 25678778